CLINICAL TRIAL: NCT00607594
Title: A Phase 2 Study of AZD0530 in Patients With Metastatic or Locally Advanced Gastric Carcinoma
Brief Title: Saracatinib in Treating Patients With Locally Advanced or Metastatic Stomach or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00188; PHL-052 (Other Grant/Funding Number: N01CM17107); CDR0000585708 (Other Grant/Funding Number: N01CM17107); PMH-PHL-052 (Other Grant/Funding Number: N01CM17107); N01CM62203 (NIH)
Record Dates: First submitted 2008-02-01; First posted 2008-02-06 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Adenocarcinoma of the Stomach; Recurrent Gastric Cancer; Stage III Gastric Cancer; Stage III Esophageal Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — saracatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (kinase inhibitor therapy) (Experimental): Patients receive saracatinib PO, at a dose of 175 mg QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Patients receive AZD0530 (saracatinib) PO QD in the absence of disease progression or unacceptable toxicity.
  Other Names: AZD0530

SUMMARY:
This phase II trial is studying how well saracatinib works in treating patients with locally advanced or metastatic stomach or gastroesophageal junction cancer. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective disease control rate (i.e., partial or complete response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or stable disease for ≥ 16 weeks) in patients with locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction treated with AZD0530 (saracatinib).

SECONDARY OBJECTIVES:

I. To assess the median time to disease progression, median overall survival, and 1-year survival rate in these patients.

II. To assess the toxicity of AZD0530 in these patients. III. To evaluate potential predictive markers by assessing pretreatment intratumoral levels of src, Y419 phospho-src (P-Src), and c-terminal src kinase (Csk) in archival tumor biopsies.

OUTLINE:

Patients receive saracatinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at least every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal junction (GEJ)

  * Tumors of the GEJ must be sub-specified as type I, II, or III using the Siewert classification
* Metastatic or locally advanced disease

  * Patients with local/regional disease only, must have unresectable disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral computed tomography (CT) scan
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Platelet count ≥ 100,000/mm³
* Leukocytes ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin > 9 g/dL
* Total bilirubin normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Urine protein creatinine ratio < 1.0 OR urine protein < 1,000 mg by 24-hour urine collection

Exclusion Criteria:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No condition that potentially impairs the ability to swallow or absorb AZD0530, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation
  * Active peptic ulcer disease
  * Short gut syndrome
  * Malabsorption syndrome of any type
  * Total or partial bowel obstruction
  * Inability to tolerate oral medications
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD0530
* No QTc prolongation (defined as a QTc interval ≥ 460 msec) or other significant electrocardiogram (ECG) abnormalities
* No poorly controlled hypertension (i.e., systolic blood pressure [BP] ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)
* No history of ischemic heart disease, including myocardial infarction
* No concurrent cardiac dysfunction including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No other concurrent uncontrolled illness, including ongoing or active infection or psychiatric illness/social situations, that would limit compliance with study requirements
* Prior chemotherapy allowed provided it was administered as part of initial curative intent therapy (i.e., neoadjuvant therapy, adjuvant therapy and/or concurrently with radiotherapy) in combination with surgery

  * At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior and no more than 1 line of palliative chemotherapy for advanced disease
* At least 4 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior major surgery and recovered
* No cytochrome 450 3A4 (CYP3A4) active agents or substances for ≥ 7 days before, during, and for ≥ 7 days after completion of study treatment
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather-Jane Au, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (5):
- Hamilton Medical Center, Dalton, Georgia, United States
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Kinase Inhibitor Therapy): Patients receive saracatinib PO QD in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  Canada | 21

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response (Defined as Partial [PR] or Complete Response [CR] by RECIST Criteria)
Description: PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. CR is defined as disappearance of all non-target lesions and normalization of tumor marker level.
Time Frame: Every 2 weeks for the first 4 weeks, and then every 4-8 weeks thereafter, for at least 16 weeks up to 37 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
participants | 0

2. Primary Outcome: Prolonged Stable Disease Rate (Defined as Stable Disease for ≥ 16 Weeks)
Time Frame: Every 2 weeks for the first 4 weeks, and then every 4-8 weeks thereafter, for at least 16 weeks up to 37 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
participants | 1

3. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions,or a measurable increase in non-target lesions, or the appearance of new lesions.
Time Frame: Up to 1 year (median, 6 month, 1-year)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
months | 1.8 [1.5 to 1.9]

4. Secondary Outcome: Progression-free Survival
Description: Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: Measured from the date of enrollment to progression, death or last contact, or last tumor assessment before the start of further anti-tumor therapy
Population: Only 17 patients were evaluable for response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 17
months | 1.8 [1.5 to 1.9]

5. Secondary Outcome: Median Survival
Description: as for outcome 4
Time Frame: Up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
months | 7.8 [3.9 to 12.2]

6. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate overall and time to progression estimates. Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. Ninety-five percent confidence intervals will be provided for estimates of interest where possible.
Time Frame: Up to 1 year (median, 6 months, and 1 year)
Population: Only 17 patients were evaluable for response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 17
months | 7.8 [3.9 to 12.2]

7. Secondary Outcome: Highest Grade Toxicity as Assessed by the National Cancer Institute (NCI) Common Toxicity Criteria Version 3.0.
Description: Toxicities will be graded using the National Cancer Institute (NCI) Common Toxicity Criteria Version 3.0.
Time Frame: Weekly during treatment
Measure: Number; unit: highest grade
Groups:
- Treatment (Kinase Inhibitor Therapy): Patients receive saracatinib PO QD in the absence of disease progression or unacceptable toxicity.
  saracatinib
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 21
highest grade | 3

8. Secondary Outcome: Patient Tolerability
Description: as for outcome 4
Time Frame: Weekly during treatment
Population: Data were not collected
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 0

9. Secondary Outcome: Association Between Correlative Markers and Clinical Outcomes
Description: as for outcome 4
Time Frame: At baseline, 6 months, and then at 1 year
Population: data were not collected
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 8/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=21)
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Confusion (Psychiatric disorders) | 1
Lung infection (Infections and infestations) | 2
Anemia (Blood and lymphatic system disorders) | 1
Death NOS (General disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Blood bilirubin increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=21)
Anemia (Blood and lymphatic system disorders) | 18
Constipation (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 14
Lymphocyte count decreased (Investigations) | 14
Anorexia (Gastrointestinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less